CLINICAL TRIAL: NCT06956963
Title: Aerobic Exercise: A Potential Rescue From the Negative Ramifications of Poor Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00006067
Record Dates: First submitted 2025-04-10; First posted 2025-05-04 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Health; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Sleep (No Intervention)
- Acute Partial Sleep Deprivation (Experimental): 30% reduction in habitual time in bed
  Interventions: Other: Partial Sleep Deprivation

INTERVENTIONS:
Other: Partial Sleep Deprivation — 30% reduction in habitual time in bed
  Other Names: Reduced Sleep
  Arms: Acute Partial Sleep Deprivation

SUMMARY:
The goal of this interventional study is to differentiate the effects of an acute partial sleep deprivation intervention on markers of cardiovascular health, cardio-autonomic function, physical and cognitive performance, as well as overall wellbeing in active vs sedentary individuals. The main aims of the project are:

* To differentiate the effects of partial sleep deprivation on central hemodynamics (i.e., central blood pressure and arterial stiffness) in active vs sedentary individuals.
* To differentiate the effects of partial sleep deprivation on physical (i.e., handgrip strength and reactive strength index) and cognitive performance (i.e., reaction time and impulse control) in active vs sedentary individuals.
* To differentiate the effects of partial sleep deprivation on overall wellbeing (i.e., cardio-autonomic function, inflammation levels, and psychological mood states) in active vs sedentary individuals.

Participants will be divided into two groups based on aerobic activity level - active or sedentary - and assessed for markers of cardiovascular health, cardio-autonomic function, physical and cognitive performance, as well as overall wellbeing before and after three days of normal sleep and three days of partially deprived sleep (i.e., 30% reduction in total time in bed).

ELIGIBILITY:
Inclusion Criteria:

* Chronically active (≥150 minutes of moderate- and/or ≥75 minutes of vigorous-intensity aerobic exercise per week for the last 3 months) OR
* Sedentary (≤60 minutes of aerobic exercise per week for the last 3 months)

Exclusion Criteria:

* Chronic, uncontrolled disease (cardiovascular, metabolic)
* Poor sleep (regularly achieving <7 hours of sleep per night)
* Musculoskeletal injury in the last 6 months
* Obese (grade II or higher)
* Pregnant

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Arterial Stiffness (i.e., carotid-femoral pulse wave velocity) | Immediately- and 3 days-post 3 days of partial sleep deprivation; Immediately- and 3 days-post 3 days of normal sleep
  Carotid-femoral pulse wave velocity measured via applanation tonometry
Central Hemodynamics | Immediately- and 3 days-post 3 days of partial sleep deprivation; Immediately- and 3 days-post 3 days of normal sleep
  Central Blood Pressure

SECONDARY OUTCOMES:
Cardio-Autonomic Function | Daily mid- and post- 3 days of partial sleep deprivation; daily mid- and post- 3 days for normal sleep
  heart rate variability
Cardio-Autonomic Function | Daily mid- and post- 3 days of partial sleep deprivation; daily mid- and post- 3 days for normal sleep
  resting heart rate
Cardio-Autonomic Function | Daily mid- and post- 3 days of partial sleep deprivation; daily mid- and post- 3 days for normal sleep
  respiration rate
Cognitive Performance | Daily mid- and post- 3 days of partial sleep deprivation; daily mid- and post- 3 days for normal sleep
  impulse control; measured via vetted smart phone application (Sway Medical; Tulsa, OK)
Cognitive Performance | Daily mid- and post- 3 days of partial sleep deprivation; daily mid- and post- 3 days for normal sleep
  reaction time; measured via vetted smart phone application (Sway Medical; Tulsa, OK)
Physical Performance | Immediately- and 3 days-post 3 days of partial sleep deprivation; Immediately- and 3 days-post 3 days of normal sleep
  hand grip strength
Physical Performance | Immediately- and 3 days-post 3 days of partial sleep deprivation; Immediately- and 3 days-post 3 days of normal sleep
  reactive strength index; scale title: reactive strength index, scale limits: 0-100, higher value is better
Inflammation | Immediately- and 3 days-post 3 days of partial sleep deprivation; Immediately- and 3 days-post 3 days of normal sleep
  CRP
Inflammation | Immediately- and 3 days-post 3 days of partial sleep deprivation; Immediately- and 3 days-post 3 days of normal sleep
  IL-6
Inflammation | Immediately- and 3 days-post 3 days of partial sleep deprivation; Immediately- and 3 days-post 3 days of normal sleep
  IL-1beta
Inflammation | Immediately- and 3 days-post 3 days of partial sleep deprivation; Immediately- and 3 days-post 3 days of normal sleep
  IL-10
Inflammation | Immediately- and 3 days-post 3 days of partial sleep deprivation; Immediately- and 3 days-post 3 days of normal sleep
  TNF-alpha

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Sciences and Medicine, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided